CLINICAL TRIAL: NCT02077920
Title: Prevention of Ventilator-Associated Pneumonia by Oropharyngeal and Subglottic Decontamination Via Bronchoscopy
Brief Title: Methods of Chlorhexidine Cleansing to Prevent Ventilator-Associated Pneumonia (VAP)
Acronym: VAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Zhuang Ma, Professor, General Hospital of Shenyang Military Region
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GHS-RCU-001
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Ventilator-associated pneumonia VAP; Chlorhexidine; Oropharyngeal decontamination; Subglottic secretion drainage
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Chlorhexidine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Chlorhexidine before intubation (Experimental): Group A: Oropharyngeal decontamination with chlorhexidine before intubation, n=48. Oral cleansing with chlorhexidine will be performed before endotracheal intubation, and every 6 hours after intubation.
  Interventions: Drug: Chlorhexidine; Device: Endotracheal tube
- Chlorhexidine after intubation (Experimental): Group B: Oropharyngeal decontamination with chlorhexidine after intubation, n=48. Oral cleansing with chlorhexidine will be performed every 6 hours after endotracheal intubation.
  Interventions: Drug: Chlorhexidine; Device: Endotracheal tube
- Subglottic secretion drainage (Experimental): Group C: Suctioning of subglottic secretions, n=48. Oral cleansing with chlorhexidine will be performed before endotracheal intubation and every 6 hours after intubation, and fiberoptic bronchoscopy-guided suctioning of subglottic secretions will be performed at 10:00 a.m. every day. The procedure will be as follows:
  1. Routine cleaning of the bronchoscope.
  2. Oral or nasal insertion of the bronchoscope (according to the decision of the attending physician based on the patient's condition). Rinsing of the subglottic region with 5-20 mL of chlorhexidine solution followed by suctioning. The rinsing procedure will be repeated 3-5 times.
  3. Routine cleaning of the bronchoscope. The patient will be monitored during all procedures.
  Interventions: Drug: Chlorhexidine; Device: Fiber bronchoscope
- 0.9% sodium chloride injection (Experimental): Group D: 0.9% sodium chloride injection, n=48. After endotracheal intubation, oral cleansing with normal saline will be performed every 6 hours.
  Interventions: Drug: 0.9% sodium chloride injection; Device: Endotracheal tube

INTERVENTIONS:
Drug: Chlorhexidine — SFDA Approval No. H21020748; Jinzhou Jiu Tai Pharmaceutical Co., Ltd., Liaoning, China
  Drug administration and preparation:
  * Drug administration: oropharyngeal rinsing and suctioning of subglottic secretions
  * Drug preparation: 0.12% chlorhexidine solution prepared with distilled water that has been sterilized by autoclaving
  Arms: Chlorhexidine after intubation; Chlorhexidine before intubation; Subglottic secretion drainage
Drug: 0.9% sodium chloride injection — SFDA Approval No. H20045252; Shenyang Zhiying Pharmaceutical Co., Ltd., Liaoning, China
  Arms: 0.9% sodium chloride injection
Device: Endotracheal tube — Type 5-10115; size 7.0 mm, 7.5 mm, or 8.0 mm; purchased from Teleflex Medical (USA).
  Arms: 0.9% sodium chloride injection; Chlorhexidine after intubation; Chlorhexidine before intubation
Device: Fiber bronchoscope — For suctioning of subglottic secretions. BF-P30 (Olympus, Japan); BF-1T20 (Olympus, Japan); or FB-18BS (Pentax, Japan).
  Arms: Subglottic secretion drainage

SUMMARY:
Ventilator-associated pneumonia (VAP) is common in patients receiving mechanical ventilation, and is associated with longer hospital stay, increased treatment costs, and higher rates of morbidity and mortality . VAP is reported to occur in 8%-67% of mechanically ventilated patients (20%-28% in most reports) and has a mortality rate of 24%-50%, which is 2-3 times the mortality rate of mechanically ventilated patients without VAP. In patients infected by multi-resistant bacteria, the mortality rate may be as high as 76%. The diagnosis, treatment, and prevention of VAP are therefore important. Strategies for preventing VAP are crucial for reducing medical costs and increasing survival rates in critically ill patients. These strategies mainly involve a semi-reclining position with the head of the bed raised to at least 30°-45°, oral care, suctioning of subglottic secretions, selective decontamination of the digestive tract, proper hand washing, avoidance or reduction of proton pump inhibitors, avoidance of excessive sedation, and control of plasma glucose levels.

At our center, VAP is mainly caused by bacterial colonization of the upper respiratory tract via aspiration. This study will compare four interventions including oropharyngeal decontamination and subglottic suctioning by bronchoscopy, with the aim of developing a prevention strategy to minimize the development of VAP during mechanical ventilation.

DETAILED DESCRIPTION:
Patients will be assessed as follows:

CABDC ABBAA BCDDA CCCDB CACBA BBABC BAAAD DCDAC CDBAA DACDD AAACB CDBCB ACCDB BBAAD BCACC DDBCA ADCAD DABCD CBAAB DDDCD AABAB ACBCD BCCBA ADCDB CBCAB CDDCA CDDDD ABCDA ABDCB CBADD ADDBA BBCCD ABBBD DCDAC BBCCB DADBB CDBDA DBBAC AC

Adverse Events:

Adverse events that occur after endotracheal intubation, mechanical ventilation, oral cleansing with chlorhexidine, and suctioning of oropharyngeal secretions by bronchoscopy will be recorded. All adverse events including laboratory abnormalities will be recorded, even if they are thought to be unrelated to medical interventions. The severity of adverse events and any correlations with experimental drugs will be carefully recorded on the case report form.

The relationships between adverse events and drug resistance will be categorized as certainly relevant, probably relevant, possibly relevant, possibly irrelevant, or certainly irrelevant. The proportions of adverse events that are categorized as certainly relevant, probably relevant, and possibly relevant will be calculated. Severe adverse events will be recorded in a table and reported to the director of the unit and the sponsor within 24 hours.

Severity Assessment:

The severity of adverse events will be categorized as mild, moderate, or severe. A mild adverse event is defined as an event with signs and symptoms that are easy to tolerate such as nausea, vomiting, or transient localized pain. A moderate adverse event is defined as an event resulting in persistent pain. A severe adverse event is defined as an event resulting in prolonged hospitalization, disability, reduced ability to work, risk of death, or congenital malformation.

The outcomes of all adverse events will be recorded. Patients who withdraw from the trial because of adverse events will be followed up until complete resolution of the events. The investigators will judge whether the adverse events are related to the administration of experimental drugs, and will record the justification for each decision.

Data Management:

Completed case report forms will be collected by the clinical coordinator and the data will be entered into the database. After checking for accuracy, the data will be locked. After unblinding, the data will be categorized according to the four groups of patients.

Statistical Analysis:

Numerical data will be described as percentages, and measurement data as mean ± standard deviation. Abnormally distributed data will be described as median and interquartile range (25th-75th percentile).

Comparisons of Baseline Data:

Numerical data will be compared between groups using the chi-square test or Fisher's exact test. Measurement data with normal distributions will be analyzed by single- or multi-factor analysis of variance. Data with high heterogeneity will be compared using a non-parametric test such as Tamhane's T2 test. Measurement data with non-normal distributions will be compared using the non-parametric Mann-Whitney U test or the Kruskal-Wallis rank sum test. Groups will be compared at baseline and at different time points after enrollment.

Comparisons of Efficacy:

Analgesic and sedative effects will be compared among groups using the Kruskal-Wallis rank sum test. For factors showing significant differences among groups, pairwise comparisons will be analyzed using the non-parametric Mann-Whitney U test. Mean values will be compared between groups using the Cochran-Mantel-Haenszel chi-square test.

Data Processing:

All statistical analyses will be performed using SAS software. Two-sided P values will be calculated. For Fisher's exact test, the P value will be calculated directly. A value of P <0.05 is considered significant, and P <0.01 is considered highly significant.

Quality Assurance:

This study will have one principal investigator, one research investigator, and four other investigators. The clinical protocol will be strictly implemented. An independent inspector will be appointed to monitor the clinical trial.

Quality Control of the Parameters Measured:

The parameters recorded will be measured according to standard operating and quality control procedures, using standard national units of measurement. Test report forms will be fully completed including the date, parameters tested, test results, and normal ranges.

Ethical Standards:

The investigators or investigator-authorized personnel will explain the benefits and risks of participating in the clinical trial to each patient, or to the patient's legal representative. Written informed consent will be obtained prior to study entry (before performance of tests and administration of drugs). The original consent forms will be stored by the investigators.

Data Retention:

The investigators will be responsible for maintaining the database and keeping the data locked for future analysis. In accordance with the principles of good clinical practice in China, the data will be kept for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are scheduled for endotracheal intubation and mechanical ventilation.

Exclusion Criteria:

* Patients who underwent endotracheal intubation or tracheotomy before study enrollment.
* Patients who underwent endotracheal intubation and mechanical ventilation within 30 days before study enrollment.
* Patients who require cardiopulmonary resuscitation.
* Patients with a history of emesis and aspiration before endotracheal intubation.
* Patients who are judged unsuitable for enrollment by clinicians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-03; Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
The incidence of Ventilator-associated Pneumonia | an expected average of 30 days
  Percentage of patients who develop VAP after endotracheal intubation

SECONDARY OUTCOMES:
Length of stay | Until discharge from hospital, an expected average of 30 days
  Number of days of hospitalization
Length of intensive care unit stay | an expected average of 30 days
  Number of days in the intensive care unit
Duration of mechanical ventilation | Until the last day of mouthpiece ventilation, an expected average of 30 days
  Influence of interventions on the duration of mechanical ventilation.
Hospital costs | During entire hospitalization, an expected average of 30 days
  Total costs incurred during hospitalization.
30-day mortality | An expected average of 30 days
  Percentage of patients who die.

OTHER OUTCOMES:
Vital signs | Before intubation, and 48 hours, 4 days, 7 days, 14 days, and 30 days after intubation
  Temperature, heart rate, blood pressure, level of consciousness
Laboratory tests | Before intubation, and 48 hours, 4 days, 7 days, 14 days, and 30 days after intubation
  White blood cell count, platelet count, throat swab culture, sputum culture, routine urinalysis, midstream urine culture, liver and kidney function tests, serum biochemistry tests, C-reactive protein level, procalcitonin level, brain natriuretic peptide level, subglottic secretion culture.
Arterial blood gas analysis | Before intubation, and 48 hours, 4 days, 7 days, 14 days, and 30 days after intubation
  pH, PO2 (mmHg), PCO2 (mmHg), lactate level (mmol/L), PO2/FiO2.
Other investigations | Before intubation, and 48 hours, 4 days, 7 days, 14 days, and 30 days after intubation
  Electrocardiography, echocardiography, chest X-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Ma, Ph.D., Principal Investigator — The General Hospital of Shenyang Military Region
Locations (1):
- The General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No